CLINICAL TRIAL: NCT05162794
Title: Is Laparoscopic Excision for Peritoneal Endometriosis Helpful or Harmful: A Double-blind, Randomized, Controlled, Three-armed Surgical Trial.
Brief Title: Is Laparoscopic Excision for Peritoneal Endometriosis Helpful or Harmful?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Aalborg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAPEX
Record Dates: First submitted 2021-11-17; First posted 2021-12-17 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2023-11

CONDITIONS: Endometriosis; Peritoneum
Keywords: Pelvic pain; Quality of life; Post-surgical neuropathic pain; Endometriosis surgery
MeSH Terms: conditions — Endometriosis; Pelvic Pain | interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Surgery (Other)
  Interventions: Other: Laparoscopy with excision; Other: Medical treatment-as-usual
- Diagnostic Surgery (Other)
  Interventions: Other: Laparoscopy without excision; Other: Medical treatment-as-usual
- No-surgery control (Other)
  Interventions: Other: Medical treatment-as-usual

INTERVENTIONS:
Other: Laparoscopy with excision — Diagnostic laparoscopy will be performed to visually confirm endometriosis in the peritoneum. Then, the relevant tissue will be excised and a histology will be performed.
  Arms: Active Surgery
Other: Laparoscopy without excision — Diagnostic laparoscopy will be performed to visually confirm endometriosis in the peritoneum. However, no tissue will be excised and histology will not be performed.
  Arms: Diagnostic Surgery
Other: Medical treatment-as-usual — Patients continue their hormonal and analgesic treatment-as-usual.

SUMMARY:
The trial seeks to test effect of laparoscopic excision of peritoneal endometriosis on pelvic pain. Data will also be gathered on quality of life and neuropathic pain. Patients will be randomized to one of three groups: 1) laparoscopy with excision of endometrial tissue, 2) laparoscopy without excision of endometrial tissue and 3) waiting list control.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years) with suspected peritoneal endometriosis undergoing elective surgery for pain relief
* Pain intensity ≥ 5 on Numeric Rating Scale (NRS) in the four weeks prior to giving consent

Exclusion Criteria:

* Other known conditions/diseases that may cause pelvic pain
* Diagnosed personality disorder, schizophrenia or treatment with anti-psychotics
* Planned pregnancy during study period
* Women who cannot read or speak Danish

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Pelvic pain measured using NRS | Change from pre-randomization to 1, 3 and 6 months post-randomization.
  Pelvic pain intensity (sensory) and unpleasantness (affective) will be measured on 11-point Numeric Rating Scales (0 = no pain to 10 = worst pain imaginable) weekly.

SECONDARY OUTCOMES:
Health-related Quality of Life measured using Endometriosis Health Profile-30 | Change from pre-randomization to 1, 3 and 6 months post-randomization.
  Quality of Life will be measured using the validated and patient-generated, endometriosis-specific questionnaire "Endometriosis Health Profile 30", consisting of 30 questions rated on Likert scales.
Neuropathic pain symptoms (patient-reported) measured using painDETECT | Change from pre-randomization to 1, 3 and 6 months post-randomization.
  Neuropathic pain symptoms (patient-reported) is measured using the validated painDETECT questionnaire.
Neuropathic pain symptoms (assessed) measured using quantitative sensory testing | Change from pre-randomization to 6 months post-randomization.
  Neuropathic pain symptoms (assessed) is measured using a quantitative sensory testing battery. Allodynia, pinprick and pressure pain thresholds are measured.
Work ability measured using "Work Ability Index" | Change from pre-randomization to 1, 3 and 6 months post-randomization.
  Work ability is measured using the "Work Ability Index" short questionnaire.
Worst pelvic pain measured using NRS | Change from pre-randomization to 1, 3 and 6 months post-randomization.
  Worst pelvic pain intensity and unpleasantness will be measured on 11-point Numeric Rating Scales (0 = no pain to 10 = worst pain imaginable) weekly.
Pain frequency measured using weekly count | Change from pre-randomization to 1, 3 and 6 months post-randomization.
  Pain frequency will be measured using a weekly count, ranging from 0 days of pain to 7 days of pain.

OTHER OUTCOMES:
Widespread pain measured using body map | Change from pre-randomization to 1, 3 and 6 months post-randomization.
  Widespread pain will be measured using a body map. At each measurement point, participants will rate the areas where they experience pain.

CONTACTS AND LOCATIONS:
Overall Officials: Axel Forman, PhD, MD, Study Director — Aarhus University, Aarhus University Hospital, Denmark; Henrik Marschall, MSc, Principal Investigator — University of Aarhus; Dorthe K Thomsen, PhD, Study Chair — University of Aarhus
Locations (5):
- Denmark (5):
  - Regional Hospital Horsens, Department of Obstetrics and Gynecology, Horsens, Central Jutland
  - Aarhus University Hospital, Department of Obstetrics and Gynecology, Aarhus N
  - Regional Hospital Herning, Department of Obstetrics and Gynecology, Herning
  - Regional Hospital Randers, Department of Obstetrics and Gynecology, Randers
  - Regional Hospital Viborg, Department of Obstetrics and Gynecology, Viborg

IPD SHARING:
Plan to Share IPD: Yes
When participant inclusion has ended, data can be shared in accordance with the ICJME guidelines, if relevant research objectives are provided. Data sharing will require approval from the Central Denmark Region and the Danish Data Protection Agency, and the requesting party shall cover any fees associated with data sharing. Requests for data can be addressed to af@clin.au.dk.

REFERENCES:
- [Derived] Marschall H, Forman A, Lunde SJ, Kesmodel US, Hansen KE, Vase L. Is laparoscopic excision for superficial peritoneal endometriosis helpful or harmful? Protocol for a double-blinded, randomised, placebo-controlled, three-armed surgical trial. BMJ Open. 2022 Nov 3;12(11):e062808. doi: 10.1136/bmjopen-2022-062808. PMID 36328387